CLINICAL TRIAL: NCT04461236
Title: Isoleucine Intake and Intermediary Metabolism in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, Associate Professor, Texas A&M University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: 2018-1486
Record Dates: First submitted 2020-06-22; First posted 2020-07-08 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Type 2 Diabetes
Keywords: Isoleucine intake
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Isoleucine (Experimental): Type 2 Diabetics randomized to isoleucine group
  Interventions: Dietary Supplement: Oral Supplement
- Placebo (Placebo Comparator): Type 2 Diabetics randomized to placebo group
  Interventions: Dietary Supplement: Placebo
- Healthy (No Intervention): gender-, age-, BMI-matched controls for baseline measurements only. No supplementation provided.

INTERVENTIONS:
Dietary Supplement: Oral Supplement — Supplement provided in capsules. Half the capsules to be taken with lunch and the other half with dinner. All supplements are commercially available.
  Arms: Isoleucine
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine the mechanism of reduced branched-chain amino acid (BCAA) oxidation to propionyl CoA and isoleucine intake can affect TCA cycle function in obese insulin resistant T2D. We will test the hypotheses that isoleucine and valine oxidation to propionyl CoA is reduced and that week long oral administration of isoleucine in T2D subjects will increase propionyl CoA and succinyl CoA production in muscle.

The secondary objectives of this study are to determine the extent to which type 2 diabetics are capable of controlling and coordinating complex patterns of force using the upper and lower limb. This line of research has functional significance as upper body coordination and fine motor control is important for many activities associated with daily living and may contribute to therapy protocols for individuals with type 2 diabetes. Functional performance via six-minute walk and balance board measurement will also be tested with and without sensory augmentation via electrical stimulation of foot. Changes in peripheral blood mononuclear cells (PBMCs) mitochondrial respiration values will also be assessed between subject types and for diabetic after the 10-day supplementation period.

DETAILED DESCRIPTION:
Defects in mitochondrial β-oxidation and branched chain amino acid (BCAA) oxidation are associated with type 2 diabetes (T2D) and other conditions such as Huntington's disease and maple syrup urine disease. Because of these defective mitochondrial pathways, production of TCA cycle intermediates can be limited and obesity worsen the condition of the disease. Interestingly, supplying precursors for the TCA cycle such as propionyl CoA can promote anaplerosis through a pathway that is independent of the defective pathway. Therefore, we hypothesize that providing oral isoleucine, a branched-chain amino acid, which is commonly used for other conditions, will promote anaplerosis by supplying the precursor, propionyl CoA for the TCA cycle intermediate succinyl CoA to muscle of T2D patients. This innovative approach is intended to improve TCA function and insulin resistance in obese T2D and could serve as a model for other nutritional interventions.

Diabetes is a growing problem worldwide and has lead to 1.5 million deaths in 2012 and it's prevalence has increased to 9% in 2014, most like related to the steep increase in obesity rates. Research has shown that a combination of increased acetyl-carnitine and reduced propionyl- and isovaleryl-carnitine and elevated blood BCAA in T2D suggests reduced BCAA oxidation to propionyl-CoA, which can cause TCA cycle a malfunction. During homeostasis, transamination of valine and isoleucine leads to α-keto-isovalerate (KIV) and α-keto-methylvalerate (KMV) production, which can be further converted to propionyl CoA and the TCA cycle intermediate succinyl-CoA. Therefore, increased valine and isoleucine transamination can promote anaplerosis and stimulate mitochondrial energetic flux. Because of this, we believe that there is a critical need to identify therapies that can be used to restore TCA function in obese T2D.

Furthermore, Type 2 diabetes causes and contributes to a variety of central nervous system (CNS) complications. CNS complications with type 2 diabetes include cognitive and motor dysfunction. There have been a number of studies investigating the association between diabetes and cognitive decline indicating deficits in psychomotor speed, executive function, memory, and attention. Research has also indicated motor deficits with complex motor skills, motor coordination, balance, and muscle strength in type 2 diabetics. However, the majority of research investigating motor dysfunction in type 2 diabetes has focused on lower body dysfunction (balance/gait) and muscular strength (grip) using gross motor control. It is not clear from the literature how type 2 diabetes influences upper body coordination and fine motor control. Chronic inflammatory states, such as obesity, congestive heart failure, diabetes, Alzheimer's disease are also linked to changes in peripheral blood mononuclear cells (PBMCs) mitochondrial respiration values]. PBMC isolation is a non-invasive way to measure mitochondrial function through high-resolution respirometry.

ELIGIBILITY:
Inclusion criteria:

* Age: 45-84 years old, inclusive
* Clinical diagnosis with type-II diabetes (Diabetics subjects only) and oral glucose lowering medication or insulin
* Stable body-weight (± 5%) for the past 3 months
* Body Mass Index (BMI): 28 kg/m2 or higher
* Subject is judged to be in satisfactory health based on medical history, physical examination, and laboratory screening evaluations.
* Ability to walk, sit down and stand up independently
* Ability to lie in supine or elevated position for up to 10 hours
* Willingness and ability to comply with the protocol

Exclusion criteria:

* Subject is expected to have surgery within one-month of screening
* Subject is currently participating or has participated in a study with an investigational compound or device within 30 days of signing the informed consent.
* Active dependence of alcohol or drugs
* Diagnosed and active treatment of Type 1 Diabetes Mellitus
* Medication: Use of substances known to influence protein metabolism: antibiotics within 3 weeks prior to the study visit, current use of corticosteroids, growth hormone, testosterone, estrogen, immunosuppressant, blood thinners, or insulin.
* Adherence to a weight loss diet.
* (Possible) pregnancy

Ages: 45 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Change in whole-body protein metabolism in type 2 diabetic obese subjects | 0, 10, 20, 40, 60, 120 ± 5 min after isotope infusion
  Change in whole-body protein synthesis rate after 10 days of isoleucine supplementation

SECONDARY OUTCOMES:
24-hour glucose levels in type 2 diabetic obese subjects | 10 days
  Blood glucose levels measured by continuous glucose monitor for 10 days of isoleucine supplementation
Group differences in fat metabolism between type 2 diabetics and non-diabetic subjects | 0, 10, 20, 40, 60, 120 ± 5 min after isotope infusion
  Whole-body production rate of glycerol in postabsorptive state
Group differences in glucose metabolism between type 2 diabetics and non-diabetic subjects | 0, 10, 20, 40, 60, 120 ± 5 min after isotope infusion
  Whole-body production rate of glucose in postabsorptive state
Changes in state of mood as measured by the Hospital Anxiety and Depression Scale (HADS) in type 2 diabetics obese subjects | postabsorptive state on study day 1 and study day 2
  Measured by a validated questionnaire on a fourteen item self-assessment scale. Seven of the items related to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 (no symptoms) and 21 (severe symptoms) for either anxiety or depression.
Changes in state of mood as measured by the Profile of Mood State (POMS) in type 2 diabetics obese subjects | postabsorptive state on study day 1 and study day 2
  A psychological distress scale to measure mood disturbance in 6 domains - fatigue-inertia, vigor-activity, tension-anxiety, depression-dejection, anger-hostility, and confusion-bewilderment. Healthy populations take 3 to 7 minutes to complete, and others may take up a bit longer.
Changes in attention and executive functions as measured by Trail Making Test (TMT) in type 2 diabetics obese subjects | postabsorptive state on study day 1 and study day 2
  In Part A, the examinee is instructed to connect a set of 25 circles with numbers as quickly as possible while maintaining accuracy. In Part B, the examinee is instructed to connect a set of 25 circles, alternating between numbers and letters, as quickly as possible while maintaining accuracy. Measures attentional resources and is a measure of the frontal lobe "executive" functions of visual search, set-switching and mental flexibility. The total time in seconds was reported for each measure.
Changes in overall cognitive abilities as measured by Montreal Cognitive Assessment (MoCA) in type 2 diabetics obese subjects | postabsorptive state on study day 1 and study day 2
  MoCa assesses several cognitive domains and is used for the screening of mild cognitive impairment. Total scores range from 0-30 with lower scores indicating decreased functioning.
Changes in attention and executive functions as measured by Brief-A in type 2 diabetics obese subjects | postabsorptive state on study day 1 and study day 2
  Brief-A is a standardized self-report that captures views of an adult's executive functions or self-regulation in his or her everyday environment.
Changes in quality of life as measured by Short Form (36) Health Survey (SF36) in type 2 diabetics obese subjects | postabsorptive state on study day 1 and study day 2
  Self administered questionnaire that measures each of the following eight health concepts: Physical Functioning (PF); Role-Physical (RP); Bodily Pain (BP); General Health (GH); Vitality (VT); Social Functioning (SF); Role-Emotional (RE); Mental Health (MH) as well as a reported Health Transition item (HT)

OTHER OUTCOMES:
Group differences in skeletal muscle strength between type 2 diabetics and non-diabetic subjects | on study day 1 (baseline)
  Skeletal muscle strength measured by handgrip and Kin-Com 1-leg test
Group differences in balance between type 2 diabetics and non-diabetic subjects | on study day 1 (baseline)
  Balance assessed by balance board test
Group differences in exercise capacity between type 2 diabetics and non-diabetic subjects | on study day 1 (baseline)
  Functional exercise capacity assessed by 6-minute walk test
Group differences in Reaction Time task between type 2 diabetics and non-diabetic subjects | on study day 1 (baseline)
  Participants attempt to match a position-time sinusoidal target with their right arm while reacting with their left arm.
Group differences in Bi-manual Coordination Task between type 2 diabetics and non-diabetic subjects | on study day 1 (baseline)
  Participants attempt to coordinate both the right and left arm to match a visual pattern.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas A&M University CTRAL, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Description to be provided: Data may be shared upon request for up to 6 years beyond completion of the trial based on methods/proposal approved by both parties' institutional review committees. Individual participant data that underlie the results of the trial may be shared after de-identification (text, tables, figures, and appendices). Additional documents available per request include: study protocol, statistical analysis plan, and informed consent. Requests should be directed to Dr. Marielle Engelen (mpkj.engelen@ctral.org).

REFERENCES:
- [Derived] Deutz LN, Wierzchowska-McNew RA, Deutz NE, Engelen MP. Reduced plasma glycine concentration in healthy and chronically diseased older adults: a marker of visceral adiposity? Am J Clin Nutr. 2024 Jun;119(6):1455-1464. doi: 10.1016/j.ajcnut.2024.04.008. Epub 2024 Apr 12. PMID 38616018
- [Derived] Wierzchowska-McNew RA, Engelen MPKJ, Thaden JJ, Ten Have GAM, Deutz NEP. Obesity- and sex-related metabolism of arginine and nitric oxide in adults. Am J Clin Nutr. 2022 Dec 19;116(6):1610-1620. doi: 10.1093/ajcn/nqac277. PMID 36166849